CLINICAL TRIAL: NCT03607162
Title: Impact of a New Sequential Approach on Antimicrobial Use in Young Children With Fever Without Source in Emergency Department
Brief Title: Impact of a PCT(Procalcitonin) Rapid Test -Based Approach on ATB (Antibiotics) Use in Children With Fever Without Source
Acronym: DIAFEVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC18_0042
Record Dates: First submitted 2018-07-10; First posted 2018-07-31 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Fever Without Source
Keywords: Bacteriemia; meningitis; Urinary tract infection; antibiotic treatment
MeSH Terms: conditions — Meningitis; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This is an open cluster randomized clinical trial with random and sequential crossover of clusters from control to intervention until all clusters are exposed. Clusters are defined as EDs.
  2 periods will be considered, one when all children will receive usual care, whatever the cluster, and a second one when, in half of the clusters, the DIAFEVER algorithm will be applied, and in the remaining clusters, children will still receive usual care.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Local usual management of FWS (pragmatic approach)
- DIAFEVER algorithm (Experimental): New DIAFEVER sequential algorithm PCT rapid test-based will be applied
  Interventions: Diagnostic Test: DIAFEVER algorithm

INTERVENTIONS:
Diagnostic Test: DIAFEVER algorithm — PCT rapid test-based predictive algorithm
  Arms: DIAFEVER algorithm

SUMMARY:
Because a newly available point-of-care test may have real interest especially for children in the Emergency Department (ED) setting, by limiting painful and stressful venipunctures and decreasing the length of stay in the ED, the investigators hypothesize that integrating this new capillary Procalcitonin (PCT) rapid test in the DIAFEVER CPR (Clinical Prediction Rules) could represent a highly valuable diagnostic tool to identify a group with low Invasive Bacterial Infection (IBI) risk and could limit unnecessary exams and antibiotic prescriptions. The aim of this present study is to demonstrate the impact of this new PCT rapid-test-based CPR on antibiotic prescription rate in young children with Fever Without Source (FWS) presenting to the ED and on morbidity and mortality

DETAILED DESCRIPTION:
This prospective multicentric randomized study will include 5000 febrile children aged six days to three years, diagnosed with fever without source, in 26 participating French and Swiss emergency departments, during a 36-month period.

During one period, all children will receive usual care. In a second period, the DIAFEVER algorithm will be applied in half of the clusters, and in the remaining clusters, children will still receive usual care.

Then in the last period of one year, all centers will apply the new PCT-based algorithm.

At day 15 after the first consultation, data concerning death, intensive care unit admission, disease-specific complications, diagnosis of bacterial infections and proportion of antibiotic treatments will be assessed by questioning parents by use of an online electronic case report form or a phone call. The endpoints will be compared between the two groups by using a mixed logistic regression model adjusted on clustering of participants within centers and period within centers.

To perform complementary studies, a biocollection will be proposed to parents when blood tests will be indicated.

ELIGIBILITY:
Inclusion Criteria:

* Febrile children aged 6 days to <36 months old presenting to an ED at their initial visit with an acute illness for a maximum of 8 days and diagnosed with a FWS defined as body temperature (measured at home or the ED) > 38°C and a physical examination by a physician without source
* Oral non-opposition will be requested from one of the parents or caregivers of the patient.
* No current antibiotic treatment or within the 48 hours before the ED presentation.
* Parental affiliation with an appropriate health insurance system
* Parents speaking French

Exclusion Criteria:

* A clear source of fever identified after a careful inspection of medical history and a physical examination
* No fever on consultation or previously subjectively assessed by parents without use of a thermometer
* Refusal of the parents to participate
* Child ≥ 36 months or < 6 days old (ie, early-onset neonatal infection)
* Ongoing ABT treatment or within the 48 hours before ED presentation
* Children with FWS who revisited the ED after their initial visit
* Participation with another interventional study involving human subjects or being in the exclusion period at the end of a previous study involving human subjects

Ages: 6 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4928 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change in antibiotics exposure | at day 15 after the first ED consultation
  Related to the superiority objective : change in antibiotics exposure based on the proportion of children who received ABT

SECONDARY OUTCOMES:
Description of the current epidemiology of FWS among children < 36 months old admitted in an ED | At inclusion visit
  The incidence of FWS among children admitted in EDs, the incidence of Severe Bacterial Infection (SBI) and IBI among the children admitted in the ED with FWS
Diagnostic value of the DIAFEVER prediction rule for SBI and IBI diagnosis | At inclusion visit
  Assessment of sensitivity, specificity, predictive values, Likelihood Ratio, of the DIAFEVER prediction rule (combining high- and intermediate-risk versus low-risk populations) considering the SBI/IBI diagnosis as the gold standard
Impact of the DIAFEVER prediction rule on median length of stay in the ED | at day 15 after the first ED consultation
Impact of the DIAFEVER prediction rule on the proportion of children with laboratory tests prescription | at day 15 after the first ED consultation
Impact of the DIAFEVER prediction rule on hospitalization rates | at day 15 after the first ED consultation
vaccine coverage of children consulting for FWS evaluated by the vaccination coverage rate (among children with FWS) | at day 15 after the first ED consultation
theoretically vaccine-preventable SBI | at day 15 after the first ED consultation
  theoretically vaccine-preventable SBI is defined as an infection with an identified serotype included in the national vaccine schedule and occurring in a child with untimely vaccination
morbidity and mortality | at day 15 after the first ED consultation
  Morbidity and mortality based on a binary composite outcome considering occurrence or not during the 15 days after discharge from the ED of one of the following events:
  * death
  * intensive care unit admission for any reason
  * disease-specific complications (ie, cerebral damage with neurologic impairment, deathless, blindness amputation, cutaneous necrosis requiring surgery, definitive renal failure etc.)
  * diagnosis of Invasive Bacterial Infection or Serious Bacterial Infection

CONTACTS AND LOCATIONS:
Locations (26):
- France (25):
  - University Hospital, Angers
  - University Hospital, Bordeaux
  - University Hospital, Brest
  - University Hospital, Caen
  - AP-HP Antoine Béclère, Clamart
  - University Hospital, Clermont-Ferrand
  - Hopital Louis Mourier, Colombes
  - Centre Hospitalier Intercommunal, Créteil
  - University Hospital, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Regional University Hospital, Lille
  - Saint Antoine Saint Vincent Hospital, Lille
  - Southern Bretagne Hospital, Lorient
  - Hospices civils de Lyon, Lyon
  - University Hospital, Montpellier
  - Regional University Hospital, Nancy
  - University Hospital, Nice
  - AP-HP Necker-Enfants Malades, Paris
  - AP-HP Robert Debré, Paris
  - Regional University Hospital, Rennes
  - CHU, Rouen
  - Saint Brieuc Hospital, Saint-Brieuc
  - Chu Saint Etienne, Saint-Etienne
  - University Hospital, Strasbourg
  - University Hospital, Toulouse
- Hopital des Enfants, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malorey D, Tavernier E, Drouard A, Vrignaud B, Bailhache M, Guyon G, Titomanlio L, Brehin C, Abalea L, Gervaix A, Basmaci R, Dubos F, Tran A, Desgranges M, Launay E, Gras-Leguen C; Diafever Study Group. Point-of-care decision rule for antibiotic prescriptions in young children with fever without source: an open cluster randomised trial. Arch Dis Child. 2025 Dec 17:archdischild-2025-329438. doi: 10.1136/archdischild-2025-329438. Online ahead of print. PMID 41407517
- [Derived] Hubert G, Launay E, Feildel Fournial C, Chauvire-Drouard A, Lorton F, Tavernier E, Giraudeau B, Gras Le Guen C. Assessment of the impact of a new sequential approach to antimicrobial use in young febrile children in the emergency department (DIAFEVERCHILD): a French prospective multicentric controlled, open, cluster-randomised, parallel-group study protocol. BMJ Open. 2020 Aug 13;10(8):e034828. doi: 10.1136/bmjopen-2019-034828. PMID 32792425